CLINICAL TRIAL: NCT06998836
Title: Exploring the Construction and Intervention Effectiveness of Dementia Prevention Education Programs for Older Adults: A Mixed-Methods Study Based on the Health Belief Model
Brief Title: Constructing and Evaluating the Effectiveness of a Community-based Older Adults Dementia Prevention Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202301106B0
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Dementia
Keywords: dementia prevention; health beliefs
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants received a structured dementia prevention education program based on focus group findings. The program included interactive sessions on dementia knowledge, risk reduction strategies, and health belief enhancement.
  Intervention(s): Dementia Prevention Education Program
  Interventions: Behavioral: Dementia prevention education
- Control Group (Active Comparator): Participants received standard health education materials in leaflet form, covering general health maintenance topics not specific to dementia.
  Intervention(s): General Health Education Leaflet
  Interventions: Other: General Health Education Leaflet

INTERVENTIONS:
Behavioral: Dementia prevention education — Dementia prevention education:A structured dementia prevention education program developed based on qualitative focus group findings. The program includes multiple interactive sessions covering dementia knowledge, health beliefs, risk reduction strategies, and motivation for preventive actions.
  Arms: Intervention Group
Other: General Health Education Leaflet — Participants received printed general health education leaflets not specifically related to dementia. The content included general wellness and health maintenance advice.
  Arms: Control Group

SUMMARY:
This study adopted a mixed-methods approach and was conducted in two exploratory phases. The first phase focused on development and involved three focus group interviews with community-dwelling older adults. These qualitative focus group discussions were used to inform the development of a dementia prevention education program based on the analysis results.

In the second phase, community-dwelling older adults were recruited to participate in the study. The experimental group received the dementia prevention education program, while the control group received general health education leaflets. Participants were assessed before the intervention, immediately after the intervention, and again three months later. The assessments measured changes in dementia-related knowledge, dementia-related worry, health beliefs, and willingness to engage in preventive actions.

This study aimed to examine the effects of the intervention on older adults' dementia knowledge, health beliefs, and willingness to undertake preventive actions.

ELIGIBILITY:
Inclusion Criteria: (1) 55 years old or above; (2) conscious and able to speak Mandarin and Taiwanese; and (3) willing to participate in this study and complete the consent form -

Exclusion Criteria:(1) diagnosed with dementia; or (2) diagnosed with severe physical or mental illness by a physician.

-

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Dementia Knowledge Score | Baseline, immediately post-intervention, 3-month follow-up
  Measured using a validated dementia knowledge questionnaire. The score reflects the participant's understanding of dementia, including symptoms, risk factors, and prevention strategies.

SECONDARY OUTCOMES:
Dementia-Related Worry Score | Baseline, immediately post-intervention, 3-month follow-up
  Measured using a standardized scale to assess the level of concern or fear participants feel toward developing dementia.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University of Science and Technology, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No